CLINICAL TRIAL: NCT03317938
Title: Unraveling Anorectal Function and Biomarker Signatures in Patients Suffering From Subtypes of Defecatory Disorders
Brief Title: Studies in Patients With Defecatory Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Giome (Other)
Responsible Party: Principal Investigator, Hans Gregersen, Professor, Giome
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017.122
Record Dates: First submitted 2017-10-03; First posted 2017-10-23 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Fecal Incontinence; Constipation
MeSH Terms: conditions — Fecal Incontinence; Constipation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fecobionics studies (Experimental)
  Interventions: Device: Fecobionics

INTERVENTIONS:
Device: Fecobionics — Fecobionics is a new device for studying defecation

SUMMARY:
Defecatory disorders like chronic constipation and faecal incontinence affect 25% of the population with rising incidence. Defecatory disorders pose a major health care burden and are poorly recognized and treated. The need for better diagnostics and therapeutics is substantial.

Current assessment of patients with constipation and faecal incontinence include endoscopic assessment to rule out intraluminal organic cause for patients' symptoms, endoanal ultrasound scan / MRI to assess patients' pelvic floor anatomy and anorectal manometry and balloon expulsion test to assess anorectal function. All tests are susceptible to measurement artifacts.

The standard technologies for anorectal assessment are anorectal manometry, balloon expulsion test and defecography. Endoluminal Functional Lumen Imaging Probe (EndoFLIP©) is a novel technology, originally used to measure the dimensions and function of a hollow organ. Anorectal manometry, balloon expulsion test, defecography, and the EndoFLIP probe will be used in the proposed studies. In addition, the proposed study intends to use a simulated feces named Fecobionics which is a device that integrates several technologies into one which will save time and reduce test variability.

In the proposed studies investigators will assess defecatory function in subgroups of Hong Kong patients suffering from chronic constipation and faecal incontinence and determine biomarkers to increase the diagnostic value of anorectal testing. Investigators will study up to 130 patients with anorectal disorders and 101 healthy control subjects. Investigators anticipate to improve diagnostics of anorectal disorders considerably and to learn about physiological mechanisms that affect defecatory efficacy.

DETAILED DESCRIPTION:
Defecatory disorders like chronic constipation and faecal incontinence affect 25% of the population with rising incidence. Defecatory disorders pose a major health care burden and are poorly recognized and treated. The need for better diagnostics and therapeutics is substantial. Currently management options for these patients are limited, partly due to the fact that control of defaecation and continence is multifactorial but also due to the fact that it is difficult to identify the exact cause of patients' incontinence. Even in healthy subjects, many aspects of defecatory mechanisms are yet not well understood.

Current assessment of patients with constipation and faecal incontinence include endoscopic assessment to rule out intraluminal organic cause for patients' symptoms, endoanal ultrasound scan / MRI to assess patients' pelvic floor anatomy and anorectal manometry and balloon expulsion test to assess anorectal function. All tests are susceptible to measurement artifacts, with a high inter-individual variation with significant overlap between healthy asymptomatic and symptomatic patients.

The standard technologies for anorectal assessment are anorectal manometry, ballon expulsion test and defecography. Endoluminal Functional Lumen Imaging Probe (EndoFLIP©) is a novel technology, originally used to measure the dimensions and function of a hollow organ. Anorectal manometry, balloon expulsion test, defecography, and the EndoFLIP probe will be used in the proposed studies. In addition, the proposed study intends to use a simulated feces named Fecobionics which is a device that integrates several technologies into one which will save time and reduce test variability. A major difference from EndoFLIP and other technologies like anorectal manometry is that the device will be defecated rather than providing static data from one location in the anal canal.

In the proposed studies investigators will assess defecatory function in subgroups of Hong Kong patients suffering from chronic constipation and faecal incontinence and determine biomarkers to increase the diagnostic value of anorectal testing. Investigators will study up to 130 patients with anorectal disorders and 101 healthy control subjects. Investigators anticipate to improve diagnostics of anorectal disorders considerably and to learn about physiological mechanisms that affect defecatory efficacy. For example, one substudy investigates the effect of posture on defecation and another substudy focuses on deferred defecation. A third study assessed defecatory parameters as a function of the stiffness of Fecobionics. Pelvic floor function will also be assessed through vaginal measurements as well as Fecobionics may be endoscopically placed in sigmoid colon. Finally, a substudy assessed intestinal parameters after insertion of Fecobionics through a stoma.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects: Asymptomatic healthy persons aged over 18 years who can give informed consent.
* CC (Chronic Constipation) Patients: Patients over 18 with history of FI for over 3months, who are able to give consent.
* FI (Fecal Incontinence) patients: Patients over 18 with history of FI for over 3months, who are able to give consent.
* Patients with a stoma who are over 18 years and able to give consent.

Exclusion Criteria:

* Healthy subjects: Persons with a history of constipation or fecal incontinence, prior abdominal surgery, medication, and diseases, especially chronic diseases that affect bowel function and defecation. Pregnant women will also be excluded.
* CC Patients: Patients, who are not willing to undergo the proposed test program and patients with prior anorectal or intestinal surgery. Pregnant women and patients with chronic dehydration and on medications like opioids will also be excluded.
* FI patients: 1) Patients who are not willing to undergo the specified tests in this study, 2) Pregnant women and 3) Patients who has had anorectal surgery or bowel resection.
* Patients with stoma: Patients, who are not willing to undergo the proposed test program and patients who have inflammation or symptoms related to the stoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Decreased anorectal pressure assessed with the Fecobionics device | 1 year
  The number of participants with low anorectal pressure during defecation

SECONDARY OUTCOMES:
Decreased anorectal mechanical stress assessed with the Fecobionics device | 1 year
  The number of participants with low anorectal mechanical stress during defecation
Decreased anorectal angle assessed with the Fecobionics device | 1 year
  The number of participants with small anorectal angle during defecation
Wave-like decrease in cross-sectional area with the Fecobionics device | 1 year
  The amount of recordings with retrograde intestinal ripples

CONTACTS AND LOCATIONS:
Locations (2):
- Hong Kong (2):
  - Prince of Wales Hospital, Hong Kong, Hong Kong
  - Department of Surgery, Prince of Wales Hospital, Hong Kong

REFERENCES:
- [Derived] Futaba K, Chen SC, Leung WW, Wong C, Mak T, Ng S, Gregersen H. Fecobionics Evaluation of Biofeedback Therapy in Patients With Fecal Incontinence. Clin Transl Gastroenterol. 2022 May 1;13(5):e00491. doi: 10.14309/ctg.0000000000000491. PMID 35363631
- [Derived] Gregersen H, Chen SC, Leung WW, Wong C, Mak T, Ng S, Daming S, Futaba K. Characterization of Patients With Obstructed Defecation and Slow Transit Constipation With a Simulated Stool. Clin Transl Gastroenterol. 2021 May 5;12(5):e00354. doi: 10.14309/ctg.0000000000000354. PMID 33949343
- [Derived] Chen SC, Futaba K, Leung WW, Wong C, Mak T, Ng S, Gregersen H. Fecobionics assessment of the effect of position on defecatory efficacy in normal subjects. Tech Coloproctol. 2021 May;25(5):559-568. doi: 10.1007/s10151-021-02439-2. Epub 2021 Mar 29. PMID 33779850
- [Derived] Gregersen H, Chen SC, Leung WW, Wong C, Mak T, Ng S, Futaba K. Novel Fecobionics Defecatory Function Testing. Clin Transl Gastroenterol. 2019 Dec;10(12):e00108. doi: 10.14309/ctg.0000000000000108. PMID 31800543